CLINICAL TRIAL: NCT00483990
Title: A Phase I, Double-blind, Stratified, Parallel Group, Placeob-controlled Study of the Safety, Tolerability and Pharmacokinetics of PSD502 (Lidocaine Prilocaine Spray) Applied to the Glans Penis up to Three Times Daily for 21 Days in Healthy Male Volunteers
Brief Title: Phase I Study of PSD502 (Lidocaine Prilocaine Spray) Applied to the Glans Penis up to Three Times a Day for 21 Days in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Plethora Solutions Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSD502-PE-003
Record Dates: First submitted 2007-06-06; First posted 2007-06-08 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-07

CONDITIONS: Healthy
Keywords: Phase I Study in healthy subjects
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PSD502

SUMMARY:
The main objective of the study is to determine the safety and tolerability of repeated application of PSD502 to the glans penis in healthy male volunteers

DETAILED DESCRIPTION:
This is a phase I, double-blind, stratified, parallel group, placebo-controlled repeat dose study in a minimum of 8 circumcised and 8 uncircumcised healthy male volunteers. Subjects will attend 2 study visits, of which 1 will be a Screening Visit (Visit 1) and the other, a consecutive 21-day treatment visit (Visit 2; Days 1-21) which commences no more than 14 days after the Screening visit. Subjects will reside in the phase I unit throughout the treatment period. The duration of each subject's participation in the study will be up to 5 weeks.

Subjects are stratified based on whether they are circumcised or uncircumcised and within each stratified group subjects are randomized to PSD502 (lidocaine prilocaine spray) or placebo in a 3:1 ratio.

Procedures during the 21 day treatment period include: visual examination of the glans penis, blood sample collection for pharmacokinetic analysis of lidocaine and prilocaine, swabbing of the glans penis for residual PSD502, vital signs and 12-lead ECG, adverse event enquiries and collection of concomitant medications. Subjects are discharged from the clinic on Day 21 following a safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Male, aged 18 years and over
* In generally good health in the opinion of the Investigator
* Willing and able to comply with all study procedures in the opinion of the Investigator

Exclusion Criteria:

* History of a significant medical condition that would preclude further study participation, in the opinion of the Investigator.
* Currently taking, or has taken within the 2 weeks prior to the Screening Visit, any concomitant medication that could confound interpretation of the safety data PSD502
* Suffering from an STD, or is positive for hepatitis B, hepatitis C, or HIV infection.
* Safety testing abnormalities at the Screening Visit, in particular liver function tests, that are indicative of a medical condition and that would preclude further participation, in the opinion of the Investigator.
* Significant abnormality of the glans penis that would preclude interpretation of the examination of the glans, or that could be worsened by use of PSD502.
* History of alcohol or drug abuse within 1 year prior to the Screening visit.
* Known drug sensitivity to amide-type local anesthetics.
* Use of an investigational (non-registered drug within 30 days of the Screening Visit.
* Unlikely to understand or be able to comply with study procedures, for any reason, in the opinion of the Investigator.
* History of Glucose-6-Phosphate Dehydrogenase (G-6-PD)deficiency or use of medications that would increase susceptibility to methemoglobinemia (e.g. anti-malarial agents).
* Use of class 1 (e.g. mexiletine, tocainide) and III (e.g. amiodarone, sotaolol)anti-arrhythmic drugs.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2007-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Safety based on: -Examination of glans penis -AEs & SAEs -Reasons for withdrawals -Use of concomitant medications -Vital signs & ECG -Urinalysis, hematology & biochemistry -Residual PSD502 on swabs

CONTACTS AND LOCATIONS:
Overall Officials: Steven F. Komjathy, MD, Principal Investigator — PRA Health Sciences
Locations (1):
- PRA International - Clinical Pharmacology Center, Lenexa, Kansas, United States